CLINICAL TRIAL: NCT07106619
Title: Evaluation of the Effect of Knee Isokinetic Strengthening Exercises on Proprioception and Balance in Stroke Patients
Brief Title: Effectiveness of Isokinetic Exercises in Proprioception for Post-stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-012
Record Dates: First submitted 2025-07-23; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: stroke rehabilitation; proprioception; isokinetic exercise
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Rehabilitation (Active Comparator): Patients will receive 15 sessions of conventional rehabilitation
  Interventions: Other: Conventional rehabilitation program
- isokinetic Exercise (Experimental): Patients will receive 15 sessions of conventional rehabilitation and 10 sessions of knee isokinetic strengthening exercise therapy for the paretic lower extremity for 3 weeks. Isokinetic strengthening exercises will be performed using Cybex 770, Humac Norm dynamometer (CSMI, Stoughton, MA, USA).
  Interventions: Device: Isokinetic Exercises; Other: Conventional rehabilitation program

INTERVENTIONS:
Device: Isokinetic Exercises — Exercises will be performed at three different angular speeds (90 ̊/sec, 5 repetitions, 5 sets; 120 ̊/sec, 8 repetitions, 5 sets; 150 ̊/sec, 10 repetitions, 5 sets).
  Arms: isokinetic Exercise
Other: Conventional rehabilitation program — Ambulation and balance exercises

SUMMARY:
Somatosensory dysfunction including the sense of movement and position, i.e. proprioception, is observed in approximately 65% of patients after stroke. Loss of muscle strength, especially in the lower extremities, and impaired proprioception lead to significant loss of function in stroke patients. In addition, recent studies have emphasised that sensory information obtained by target-oriented exercises plays an important role in neuroplasticity and proprioception is an important element. The aim of this study was to evaluate the effect of knee isokinetic muscle strengthening exercises on proprioception and balance in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months and no more than 1 year must have passed since the date of the incident
* Be between 35 and 75 years of age
* Manual muscle testing of the affected lower extremity shows at least 3 in ankle dorsiflexion and knee extension
* No limitation in passive joint range of motion in the lower extremity
* Mini mental test score > 23

Exclusion Criteria:

* Presence of spasticity according to the modified Ashworth scale > 1+
* Presence of neurological disease other than stroke
* Presence of other medical conditions that may cause sensorimotor dysfunction in the lower extremities (e.g., diabetic polyneuropathy)
* Presence of orthopaedic problems affecting lower extremity function
* Previous history of stroke or ischaemic attack
* Poor general health status (e.g. severe heart failure, COPD)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proprioception assessment with isokinetic test device | before treatment and at the 3rd week of treatment

SECONDARY OUTCOMES:
Berg scale | Before treatment and at 3rd week of treatment
Time up and Go Test | Before treatment and at the 3rd week of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)